CLINICAL TRIAL: NCT05139667
Title: Evaluation of Mucoadhesive Tacrolimus Patch on Caspase-3 Inducing Apoptosis in Oral Lichen Planus ( A Randomized Controlled Clinical Trial With Immunohistochemical Analysis)
Brief Title: Evaluation of Mucoadhesive Tacrolimus Patch on Caspase-3 Inducing Apoptosis in Oral Lichen Planus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Dawoud, assistant lecturer of oral medicine and diagnosis, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECD123
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Adrenal Cortex Hormones; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: treatment of oral lichen planus
Who Masked: Outcomes Assessor
Masking Description: oral lichen planus
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tacrolimus/corticosteroid (Experimental): topical steroids ( triamcinolone acetonide 0.1 %), tacrolimus paste and tacrolimus patch
  Interventions: Drug: Corticosteroid Topical
- corticosteroids (Active Comparator): topical corticosteroid
  Interventions: Drug: Corticosteroid Topical
- tacrolimus (Active Comparator): topical tacrolimus patch and tacrolimus paste
  Interventions: Drug: Corticosteroid Topical

INTERVENTIONS:
Drug: Corticosteroid Topical — topical tacrolimus and corticosteroids
  Other Names: tacrolimus paste and patch topical

SUMMARY:
tacrolimus has been widely used as an immunosuppressant. the objective of this study was to evaluate the clinical efficacy of tacrolimus 0.1 % in muco adhesive patch compared to tacrolimus or corticosteroids in paste forms for symptomatic oral lichen planus, and to investigate the effect of topical tacrolimus or corticosteroids on the expression of caspase-3 in oral lichen planus as an early marker of apoptosis using immunohistochemically analysis

DETAILED DESCRIPTION:
thirty patients with erosive or atrophic OLP were randomly assigned into three equal groups to receive topical steroid ( triamcinolone acetonide 0.1%), four times per day ( Group 1), tacrolimus paste 0.1% four times per day ( Group 2) , and tacrolimus patch 2 times per day ( Group 3). all groups are given treatment for 8 weeks and 4 weeks follow up period without treatment. Photographs of the most severe lesion were taken ( marker lesion ) in each patient and analyzed for total ulcerative area (TUA), total atrophic area (TAA). patients were also assessed using clinical scores (CS) and visual analogue scale (VAS). pre treatment and post treatment specimens were immunohistochemically stained to detect expression of caspase-3.

ELIGIBILITY:
Inclusion Criteria:

* clinically and histologically proven painful bullous/erosive or atrophic forms of OLP

Exclusion Criteria:

* lichenoid lesions smoking systemic conditions pregnancy or breast feeding known hypersnstivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
clinical score | change from baseline at 12 weeks
  "0" represnted no lesion/normal mucosa, "1" mild white stria / no erythematous area

SECONDARY OUTCOMES:
caspase-3 | change from base line at 8 weeks
  caspase-3 cells count in immunostained section

CONTACTS AND LOCATIONS:
Locations (1):
- Noha Dawoud, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim SS, Ragy NI, Nagy NA, El-Kammar H, Elbakry AM, Ezzatt OM. Evaluation of muco-adhesive tacrolimus patch on caspase-3 induced apoptosis in oral lichen planus: a randomized clinical trial. BMC Oral Health. 2023 Feb 14;23(1):99. doi: 10.1186/s12903-023-02803-8. PMID 36788511